CLINICAL TRIAL: NCT06270719
Title: A Long-term Multicenter Prospective Observational Study Evaluating the Comparative Effectiveness and Safety of Sarepta Gene Transfer Therapy vs. Standard of Care in Participants With Duchenne Muscular Dystrophy Under Conditions of Routine Clinical Practice
Brief Title: An Observational Study Comparing Delandistrogene Moxeparvovec With Standard of Care in Participants With Duchenne Muscular Dystrophy
Acronym: ENDURE
Status: Enrolling by invitation | Type: Observational
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SRP-9001-401
Record Dates: First submitted 2024-01-24; First posted 2024-02-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Observational; Standard of Care; Phase 4
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Delandistrogene Moxeparvovec: Participants in Cohort 1 will have a plan for prescription of delandistrogene moxeparvovec commercially as part of clinical care prior to entry into this study.
  Cohort 1a includes participants who are ambulatory and aged 4 years or greater at baseline prescribed delandistrogene moxeparvovec commercially and recruited by treating physicians before infusion is administered.
  Cohort 1b includes non-ambulatory DMD participants aged 4 years or greater at baseline prescribed delandistrogene moxeparvovec commercially and recruited by treating physicians before infusion is administered.
  Interventions: Genetic: Delandistrogene Moxeparvovec
- Cohort 2: Standard of Care: Cohort 2 includes ambulatory DMD participants aged 4 years or greater at baseline unexposed to DMD gene therapy and receiving standard of care therapy (chronic glucocorticoid treatment) at study entry with or without baseline use of other DMD approved therapies.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Genetic: Delandistrogene Moxeparvovec — No study medication will be provided by the sponsor during this study.
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
  Groups: Cohort 1: Delandistrogene Moxeparvovec
Drug: Standard of Care — No study medication will be provided by the sponsor during this study.
  Other Names: Chronic glucocorticoid treatment
  Groups: Cohort 2: Standard of Care

SUMMARY:
This is a multicenter, prospective, observational Phase 4 study in the United States. The study is designed to collect both medical history and prospective data on Duchenne muscular dystrophy (DMD) treatment outcomes in participants receiving delandistrogene moxeparvovec as part of clinical care, compared to participants with DMD receiving or prescribed to start chronic glucocorticoid treatment at baseline in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Has a definitive diagnosis of DMD prior to Screening based on documentation of clinical findings and confirmatory genetic testing.
* Is currently receiving or has been prescribed to start chronic glucocorticoid therapy at the time of this observational study enrollment.

A participant recruited to Cohorts 1a or 2:

* Is at least 4 years of age at the time of enrollment.
* Is ambulatory per protocol specified criteria.

A participant recruited to Cohort 1b:

- Is non-ambulatory per protocol-specified criteria.

For Delandistrogene Moxeparvovec-treated Participants:

- Will be initiating usual care treatment with delandistrogene moxeparvovec at the time of study enrollment.

For Comparators:

- Is unexposed to DMD gene therapy at the time of study enrollment.

Exclusion Criteria:

* Has any deletion of exon 8 and/or exon 9 in the DMD gene.
* Is currently participating in any DMD interventional study at the time of this observational study enrollment.
* Has a medical condition or confounding circumstances (for example, prior traumatic limitation for mobility or significant behavioral comorbidity) that, in the opinion of the Investigator, might compromise:

  * The participant's ability to comply with the protocol-required procedures,
  * The participant's wellbeing or safety, and/or
  * The clinical interpretability of the data collected from the participant.

Other inclusion/exclusion criteria may apply.

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DMD participants within each prescriber's practice who either (1) have been prescribed delandistrogene moxeparvovec or (2) are receiving or have been prescribed to begin chronic glucocorticoid therapy in routine clinical practice, and who meet the study eligibility criteria, will be invited to enroll into the study and will be followed according to the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Time to Walk/Run 10 Meters (10MWR) (Calculated Velocity) at Month 12 | Baseline, Month 12

SECONDARY OUTCOMES:
Time to Rise From Floor (Supine to Stand) | Up to 10 years
Loss of Ambulation (LOA) | Up to 10 years
Performance of Upper Limb (PUL) Version 2.0 Entry Item A Score | Up to 10 years
Patient-reported Outcomes Measurement Information (PROMIS) Domain Scores of Mobility, Upper Extremity and Fatigue | Up to 10 years
Pulmonary Function, as Measured by Forced Vital Capacity (FVC) (% Predicted) | Up to 10 years
Cardiac Function, Including Left Ventricular Ejection Fraction (LVEF) as Measured by Echocardiogram (ECHO) | Up to 10 years
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to 10 years
Time to Walk/Run 10 Meters (Calculated Velocity) | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles - PIN, Los Angeles, California
  - University of Colorado - PPDS, Aurora, Colorado
  - Connecticut Children's Medical Center - Hartford, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital - Orlando, Orlando, Florida
  - All Children's Research Institute, Inc, St. Petersburg, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana Clinical and Translational Science Institute, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Duke Lenox Baker Children's Hospital, Durham, North Carolina
  - Childrens Hospital Medical Center of Akron, Akron, Ohio
  - OHSU Healthcare (Oregon Health and Science University), Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Hospital, Fort Worth, Texas
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - The Board of Regents of the University of Wisconsin, Madison, Wisconsin
  - The Medical College of Wisconsin, Milwaukee, Wisconsin